CLINICAL TRIAL: NCT06208683
Title: The Immunogenicity and Safety of the Booster Doses of a Live-attenuated Mumps Vaccine Administrated Alone and Concomitantly With a Quadrivalent Inactivated Influenza Vaccine in Junior High School Students
Brief Title: The Immunogenicity and Safety of the Booster Doses of a Live-attenuated Mumps Vaccine in Junior High School Students
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO-MUM-MA4001-SN
Record Dates: First submitted 2023-11-23; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2023-11

CONDITIONS: Mumps; Influenza
MeSH Terms: conditions — Mumps; Influenza, Human | interventions — Mumps Vaccine; Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1MCV: MV (Experimental): 100 students with a history of 1 dose of MCV will receive 1 dose of MV.
  Interventions: Biological: Mumps vaccine, Live (MV)
- 1MCV: QIV (Experimental): 100 students with a history of 1 dose of MCV will receive 1 dose of QIV.
  Interventions: Biological: Influenza Vaccine, inactivated, quadrivlent(QIV)
- 1MCV: MV +QIV (Experimental): 100 students with a history of 1 dose of MCV will receive 1 dose of MV and 1 dose of QIV simultaneously.
  Interventions: Biological: Mumps vaccine, Live (MV); Biological: Influenza Vaccine, inactivated, quadrivlent(QIV)
- 2MCV: MV (Experimental): 100 students with a history of 2 dose of MCV will receive 1 dose of MV.
  Interventions: Biological: Mumps vaccine, Live (MV)

INTERVENTIONS:
Biological: Mumps vaccine, Live (MV) — 0.5mL per dose,containing ≥3.7 lg CCID50 live mumps virus
  Arms: 1MCV: MV; 1MCV: MV +QIV; 2MCV: MV
Biological: Influenza Vaccine, inactivated, quadrivlent(QIV) — 0.5mL per dose, containing 4 strains of influenza virus recommended by the WHO, 15ug of each strain.
  Arms: 1MCV: MV +QIV; 1MCV: QIV

SUMMARY:
This study is a randomized, controlled, open-label phase Ⅳ clinical trial of a live attenuated mumps vaccine manufactured by Sinovac (Dalian) Vaccine Technology Co., Ltd. The purpose of this study is to evaluate the immunogenicity and safety of the booster doses of a mumps vaccine administrated alone and concomitantly with a quadrivalent inactivated influenza vaccine in healthy junior high school students. And the cross-neutralization of mumps vaccine immune serum and mumps virus strains

DETAILED DESCRIPTION:
This study is an open-lable, randomised, controlled phase Ⅳ clinical trial in healthy junior high school students to the immunogenicity and safety of the booster doses of a mumps vaccine (MV) administrated alone and concomitantly with a quadrivalent influenza vaccine (QIV) in healthy junior high school students. The experimental vaccine was manufactured by Sinovac (Dalian) Vaccine Technology Co., Ltd. A total of 400 healthy students will be enrolled, including 300 students who have received one dose of mumps-containing vaccine (MCV) before vaccination, and 100 students who have received two doses of mumps-containing vaccine before vaccination. 300 students with a history of 1 dose of MCV will be randomly divided into 3 groups in a ratio of 1:1:1, and will receive 1 dose of MV alone, 1 dose of QIV alone, or 1 dose of MV and 1 dose of QIV simultaneously. Students with a history of 2 doses of MCV received 1 dose of MV alone. Blood samples were collected before and 30 days after vaccination. Pre-vaccination blood samples were used to detect antibody levels of measles, mumps, influenza and varicella, and post-vaccination blood samples were used to detect mumps antibodies and/or influenza antibodies corresponding to the vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Healthy junior high school students;
* subjects and/or guardians who can understand and voluntarily sign the informed consent form (For subjects aged 8-17 years, both subjects and guardians need to sign the informed consent form)
* Provision of valid identification.;
* History of 1 or 2 doses of mumps-containing vaccine;

Exclusion Criteria:

* History of mumps or have completed 3 doses of mumps-containing vaccine;
* Receipt of the current seasonal influenza vaccine (except subjects in Arm 4)
* History of asthma or allergy to the vaccine or vaccine components, or serious adverse reactions to the vaccine, such as urticaria, dyspnea,and angioedema;
* Congenital malformations or developmental disorders, genetic defects, severe malnutrition;
* Autoimmune disease (such as systemic lupus erythematosus) or a state of immunodeficiency / immunosuppression (such as AIDS, after organ transplantation);
* Severe chronic diseases, severe cardiovascular diseases, hypertension and diabetes that cannot be controlled by drugs, liver or kidney diseases, malignant tumors, etc.;
* Severe neurological disease (epilepsy, convulsions or convulsions) or mental illness;
* Thyroid disease or history of thyroidectomy, asplenia, functional asplenia, any condition resulting in asplenia or splenectomy;
* Abnormal coagulation function diagnosed by a doctor (such as coagulation factor deficiency, coagulation disease, platelet abnormality) or obvious bruising or coagulation disorder;
* Immunosuppressive therapy, cytotoxic therapy, inhaled corticosteroids (excluding corticosteroid spray therapy for allergic rhinitis, topical corticosteroid therapy for acute uncomplicated dermatitis) within the past 6 months;
* Receipt of blood products in the past 3 months;
* Receipt of other investigational drugs in the past 30 days;
* Receipt of attenuated live vaccines in the past 28 days;
* Receipt of inactivated or subunit vaccines in the past 7 days;
* Onset of various acute or chronic diseases within 7 days prior to the study;
* Axillary temperature >37.0°C;
* Participation in other clinical trials before enrollment and during the follow-up period, or a plan to participate in other clinical trials within 3 months.
* Any other factors that are unsuitable for participating in this clinical trial according to the investigator's judgment

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2023-11-04 (Actual); Primary Completion 2024-02-02 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Geometric mean concentrations (GMCs) of mumps antibody | 30 days after the vaccination of MV
  GMC s of mumps antibody 30 days after the vaccination of MV

SECONDARY OUTCOMES:
Geometric mean increases (GMIs) of mumps antibody | 30 days after the vaccination of MV
  Geometric mean increases (GMIs) of mumps antibody 30 days after the vaccination of MV
Seroconversion rate of mumps antibody | 30 days after the vaccination of MV
  Seroconversion rate of mumps antibody 30 days after the vaccination of MV
Seropositivity rate of mumps antibody | 30 days after the vaccination of MV
  Seropositivity rate of mumps antibody 30 days after the vaccination of MV
Geometric mean titers (GMTs) of influenza antibody | 30 days after the vaccination of QIV
  Geometric mean titers (GMTs) of influenza antibody 30 days after the vaccination of QIV
Geometric mean increases (GMIs) of influenza antibody | 30 days after the vaccination of QIV
  Geometric mean increases (GMIs) of influenza antibody 30 days after the vaccination of QIV
Seroconversion rate of influenza antibody | 30 days after the vaccination of QIV
  Seroconversion rate of influenza antibody 30 days after the vaccination of QIV
Seropositivity rate of influenza antibody | 30 days after the vaccination of QIV
  Seropositivity rate of influenza antibody 30 days after the vaccination of QIV
Geometric mean concentrations (GMCs) of mumps antibody 30 days after the simultaneous vaccination of MV and QIV | 30 days after the simultaneous vaccination of MV and QIV
  Geometric mean concentrations (GMCs) of mumps antibody
Geometric mean titers (GMTs) of influenza antibody 30 days after the simultaneous vaccination of MV and QIV | 30 days after the simultaneous vaccination of MV and QIV
  Geometric mean titers (GMTs) of influenza antibody
Geometric mean increases (GMIs) of mumps antibody and influenza antibody | 30 days after the simultaneous vaccination of MV and QIV
  Geometric mean increases (GMIs) of mumps antibody and influenza antibody 30 days after the simultaneous vaccination of MV and QIV
Seroconversion rate of mumps antibody and influenza antibody | 30 days after the simultaneous vaccination of MV and QIV
  Seroconversion rate of mumps antibody and influenza antibody 30 days after the simultaneous vaccination of MV and QIV
Seropositivity rate of mumps antibody and influenza antibody | 30 days after the simultaneous vaccination of MV and QIV
  Seropositivity rate of mumps antibody and influenza antibody 30 days after the simultaneous vaccination of MV and QIV
The incidence of adverse reactions 0-7 days after vaccination | 0-7 days after vaccination
  The incidence of adverse reactions 0-7 days after vaccination
The incidence of adverse reactions 0-14 days after vaccination | 0-14 days after vaccination
  The incidence of adverse reactions 0-14 days after vaccination
The incidence of adverse reactions 0-30 days after vaccination | 0-30 days after vaccination
  The incidence of adverse reactions 0-30 days after vaccination
Geometric mean concentrations (GMCs) of measles antibody before vaccination | before vaccination
  Geometric mean concentrations (GMCs) of measles antibody before vaccination
Geometric mean concentrations (GMCs) of rubella antibody before vaccination | before vaccination
  Geometric mean concentrations (GMCs) of rubella antibody before vaccination
Geometric mean titers (GMTs) of varicella-zostor antibody before vaccination | before vaccination
  Geometric mean titers (GMTs) of varicella-zostor antibody before vaccination
Geometric mean concentrations (GMCs) of mumps antibody before vaccination | before vaccination
  Geometric mean concentrations (GMCs) of mumps antibody before vaccination
Geometric mean titers (GMTs) of influenza antibody before vaccination | before vaccination
  Geometric mean titers (GMTs) of influenza antibody before vaccination
Seropositivity rate of measles antibody before vaccination | before vaccination
  Seropositivity rate of measles antibody before vaccination
Seropositivity rate of rubella antibody before vaccination | before vaccination
  Seropositivity rate of rubella antibody before vaccination
Seropositivity rate of varicella-zostor antibody before vaccination | before vaccination
  Seropositivity rate of varicella-zostor antibody before vaccination
Seropositivity rate of mumps antibody before vaccination | before vaccination
  Seropositivity rate of mumps antibody before vaccination
Seropositivity rate of influenza antibody before vaccination | before vaccination
  Seropositivity rate of influenza antibody before vaccination
Cross-neutralizing antibody titer of mumps vaccine | 30 days after the vaccination of MV alone or simultaneously with QIV
  Cross-neutralizing antibody titer of mumps vaccine against different genotypes of mumps virus

CONTACTS AND LOCATIONS:
Overall Officials: Weijun Hu, Master, Principal Investigator — Shaanxi Provincial Center for Disease Prevention and Control
Locations (3):
- China (3):
  - Qindu Distric Center for Disease Prevention and Control, Xianyang, Shaanxi
  - Xingping Center for Disease Prevention and Control, Xianyang, Shaanxi
  - Yuyang Distict Center for Disease Prevention and Control, Yulin, Shaanxi